CLINICAL TRIAL: NCT07064772
Title: The Immediate Effects of First Rib Mobilization on Pain and Range of Motion in Patients With Shoulder Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrews University (Other)
Collaborators: Lebanon Valley College (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-095
Record Dates: First submitted 2025-07-07; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Shoulder Pain
Keywords: Manual Therapy; Physical Therapy; First Rib; Joint Mobilization; Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Rib Mobilization Group (Experimental): Participants in this arm will be randomly assigned to receive a first rib mobilization on their affected side of shoulder pain by a licensed physical therapist.
  Interventions: Other: First Rib Mobilization
- Sham Mobilization (Sham Comparator): Participants in this arm will be randomly assigned to receive a sham mobilization to the region of the first rib on their affected side of shoulder pain by a licensed physical therapist.
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Other: First Rib Mobilization — Participants in the mobilization group will receive either a seated or supine three stage progressive muscle energy technique (MET) plus a singular high-velocity, low-amplitude thrust (HVLAT) mobilization technique directed to their first rib on their symptomatic side based on the discretion of the treating physical therapist.
  Arms: First Rib Mobilization Group
Other: Sham Comparator — Participants in the sham mobilization (control) group will be placed in a supine, hook-lying position identical to the mobilization group; however, they will be instructed to inhale and exhale 3 times using diaphragmatic breathing (avoiding upper chest recruitment) as the physical therapist gently rests his or her hand over the area of the upper trapezius muscle just proximal to the first rib to simulate a sham mobilization hand placement. Therefore, physical therapists will not use any significant compressive force to the musculature, perform any tactile cueing for upper chest breathing, perform any mobilizations, nor perform any HVLAT techniques to participants in the sham mobilization group.
  Arms: Sham Mobilization

SUMMARY:
The purpose of this clinical trial is to examine whether one session of a specific manual physical therapy technique, known as first rib mobilization, can lead to immediate improvements in pain and movement in individuals with shoulder pain. We hypothesize that this single treatment will result in reduced pain and increased ability to move the shoulder and neck. Researchers will compare first rib mobilization to a sham mobilization (a look-alike hands-on position that does not mobilize the first rib) to see if first rib mobilization works to immediately reduce pain and improve movement in patients with shoulder pain.

Participants will receive first rib mobilization or a sham mobilization during a single session of physical therapy and will receive pre and post intervention measurements of their pain levels and neck and shoulder range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women
* Ages 18-75 years old
* Attending physical therapy
* Primary complaint of shoulder pain
* Pain intensity >3/10 on the Numeric Pain Rating Scale (NPRS)
* A Quick Disabilities of the Arm, Shoulder, and Hand Questionnaire (Quick DASH) score greater than 16% impaired

Exclusion Criteria:

* Previous shoulder or neck surgery
* Clinical signs of a full rotator cuff tear (positive drop arm test)
* Having positive MRI findings of a complete rotator cuff tear
* Having a positive Spurling's test
* Having a steroid injection in the cervical spine and/or shoulder in the last two months
* Having any red flags (history of cancer, upper motor neuron disorder, fractures, osteoporosis, acute inflammatory process)
* Expressing fear/anxiety related to receiving manual therapy treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-07-14 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Range of motion | Cervical and shoulder active range of motion will be assessed in participants in both groups at baseline and immediately following the intervention
  Cervical and Shoulder active range of motion
Pain Intensity | Change in pain intensity from baseline to immediately following intervention in both groups
  Pain Intensity will be assessed via the Numeric Pain Rating Scale (NPRS). On this scale, zero is equivalent to no pain and 10 indicates the worst possible pain.

SECONDARY OUTCOMES:
Global Rating of Change | This will be administered to participants in both groups immediately after intervention
  The GROC is a single-item measure that captures a patient's perceived change in their condition over time. It uses a 15-point scale ranging from -7 ("a very great deal worse") to +7 ("a very great deal better"), with 0 indicating "no change."

CONTACTS AND LOCATIONS:
Locations (1):
- Lebanon Valley College, Annville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) Sharing Statement
  Plan to Share IPD: Yes
  Description: Deidentified individual participant data (IPD) that underlie the results of this study will be shared.
  Time Frame: Data will be available beginning 3 months following publication and will remain available for 5 years.
  Access Criteria: Access will be granted to qualified researchers with a methodologically sound proposal, subject to approval by the study investigators. Proposals should be submitted to the corresponding author.
  Data Access Contact Information: Joseph R. Hribick, hribick@andrews.edu
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available beginning 3 months following publication and will remain available for 5 years.
Access Criteria: Access will be granted to qualified researchers with a methodologically sound proposal, subject to approval by the study investigators. Proposals should be submitted to the corresponding author.